CLINICAL TRIAL: NCT03987997
Title: Bed Rest and Muscle Strength in Resuscitation Patients: Interest in the Early Association of NEMS With Cyclo-ergometer Mobilization
Brief Title: Bed Rest and Muscle Strength in ICU: Interest in the Early Association of NEMS With Cyclo-ergometer Mobilization
Acronym: AFMPR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2016RC02; 2018-A01330-55 (Registry Identifier: IDRCB)
Record Dates: First submitted 2019-05-13; First posted 2019-06-17 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Weakness, Muscle
Keywords: Intensive Care Units; Critical Illness; Rehabilitation; Muscle atrophy; Muscle weakness; Cyclo-ergometer; Electrical muscle stimulation
MeSH Terms: conditions — Muscle Weakness; Critical Illness; Muscular Atrophy

STUDY DESIGN:
Intervention Model Description: Leg with electrical muscle stimulation and cycling versus leg with cycling only
Who Masked: Outcomes Assessor
Masking Description: Only one leg receives the electrical muscle stimulation, the leg which receives the electrical stimulation is randomized. An outcome assessor assess the outcome blindly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Association electrical muscle stimulation with cyclo-ergometer (Active Comparator): Randomized leg with receive electrical muscle stimulation of the quadriceps in addition to early mobilization of lower limbs with cyclo-ergometer.
  Interventions: Device: Early association of electrical muscle stimulation with cyclo-ergometer
- Cyclo-ergometer only (Other): This control group correspond to the leg which don't receive electrical muscle stimulation (as usually supported)
  Interventions: Device: Early association of electrical muscle stimulation with cyclo-ergometer

INTERVENTIONS:
Device: Early association of electrical muscle stimulation with cyclo-ergometer — Early electrical muscle stimulation in patients usually mobilized with cyclo-ergometer in ICU.

SUMMARY:
Muscles atrophy and weakness are common in intensive care units, their origin is multifactorial. Passive then active mobilization with cyclo-ergometer have shown to improve functional abilities and limit muscle weakness among intensive care unit patients. Electrical muscle stimulation should limit the atrophy and muscle weakness in intensive care unit associated with early mobilization.

This study aims to compare the association early cyclo-ergometer mobilization with electrical muscle stimulation versus cyclo-ergometer mobilization only to prevent muscle atrophy and weakness in intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Patient affiliated to a social security scheme
* Patient hospitalized in intensive care unit for medical or surgical reasons, under assisted ventilation (invasive, non-invasive ventilation or oxygen-therapy at high speed via the Optiflow(r) system delivering a flow between 30 and 60 L.min and a FiO2 between 30 and 100%)
* State of the patient deemed stable buy the doctor responsible for the care and allowing the action of the physiotherapist (acts on medical prescription)
* Age more than 18 years old (major patient) and less than 75 years old
* Duration of mechanical ventilation (invasive or not) less than or equal to 72 hours at the beginning of the inclusion
* Predicable duration of stay greater than or equal to 3 days

Exclusion Criteria:

* Impossibility to know the consent of the patient, his legal representative or the person of trust
* Patient under safeguard of justice, tutorship or curatorship
* Legionnaire not rectified
* Cardiac stimulator or defibrillator
* Cardiorespiratory state clinically not compatible withe early mobilization
* Neurological problems: intracranial pressure > 20 mmHg, presence of ICU acquired neuropathy, pre-existing diagnosis of neuromuscular disease (MS, ALS...), acute stroke, epilepsy
* Orthopedic problems: even partial amputation of a lower limb, unstable fracture, suspicion of fracture, non-fixed spinal cord injury, use of a technique that does not allow to comply with postoperative surgical instructions (range of motion, discharge...), untreated deep vein thrombosis, traumatic sequelae to the origin of disabling manifest muscle weakness of a lower limb at admission
* Dermatological problems: severe lesions or complex dressing in the lower limbs
* Morphological criteria : size < 1.5m, BMI > 35
* Confirmed psychiatric illness or severe agitation
* Abdominal surgery without protection by compression belt (medical prescription), or too fragile (medical opinion)
* Pregnant or lactating women (postpartum is not an exclusion criterion)
* Patients over 75 years old
* Hemiplegia / sequential hemiparesis
* Impossibility to practice electrostimulation on at least one lower limb (manifest muscle weakness of a lower limb at admission (e. g. related to a traumatic sequelae)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2018-08-09 (Actual); Primary Completion 2021-11-26 (Estimated); Study Completion 2021-12-26 (Estimated)

PRIMARY OUTCOMES:
Change of muscle mass of quadriceps assessed with ultrasonography | at day 0, then every 7 days (+/- 2 days) until ICU discharge (at least 6 months)
  Muscle mass of quadriceps assessed by ultrasonography. The member who receives the cyclo-ergometer mobilization alone serves as a control for the member who receives the mobilization by cyclo-ergometer and electrical muscle stimulation

SECONDARY OUTCOMES:
Change of muscle strength of lower limb assessed by dynamometry | at day 0, then every 7 days (+/- 2 days) until ICU discharge (at least 6 months)
  Muscle strength of lower limb assessed by dynamometry. The member who receives the cyclo-ergometer mobilization alone serves as a control for the member who receives the mobilization by cyclo-ergometer and electrical muscle stimulation
Change of pedalling symmetry right/left | at day 0, then every 7 days (+/- 2 days) until ICU discharge (at least 6 months)
  Assessed with the cyclo-ergometer associated pic torque
Change of power variation of lower limb | at day 0, then every 7 days (+/- 2 days) until ICU discharge (at least 6 months)
  Power variation of lower limb assessed with cyclo-ergometer
Change of work variation of lower limb | Every cyclo-ergometer session, 5 days on 7 (at least 6 months)
  Work variation of lower limb assessed with cyclo-ergometer

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital d'intruction des armées Clermont-Tonnerre, Brest, France

IPD SHARING:
Plan to Share IPD: No